CLINICAL TRIAL: NCT05785637
Title: Initiation of Polygraphy for Neuromuscular Disease Patients Under Non-invasive Mechanical Ventilation
Brief Title: Polygraphy at Home for Neuromuscular Patients Under Non-invasive Mechanical Ventilation
Acronym: HPforNIV
Status: Recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Association Française contre les Myopathies (AFM), Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP230176; 2022-A01925-38 (Registry Identifier: IDRCB)
Record Dates: First submitted 2023-03-14; First posted 2023-03-27 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Neuromuscular Diseases
Keywords: Neuromuscular Diseases; Polygraphy
MeSH Terms: conditions — Neuromuscular Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Initiation a non-invasive ventilation at night: Neuromuscular patients with chronic respiratory failure who initiate a non-invasive ventilation at night.
  Interventions: Procedure: Polygraphy diagnostic at home

INTERVENTIONS:
Procedure: Polygraphy diagnostic at home — Polygraphy diagnostic at home for patients under non-invasive mechanical ventilation.

SUMMARY:
The primary objective of the study is to evaluate the feasibility, the quality and the utility of a polygraphic control at home in order to appreciate the efficacy of the night time non-invasive ventilation (allowing to optimize the ventilator settings when the results are not satisfactory).

ELIGIBILITY:
Inclusion Criteria:

* Patient ≥ 18 years;
* Patient with chronic respiratory insufficiency has just been posed non-invasive ventilation (NIV) in the hospital, according to the latest international recommendations ;
* Affiliation to the social security scheme;
* Patient has signed the informed consent form to participate to the study.

Exclusion Criteria:

* Patient refusal;
* Patient under guardianship;
* Patient under AME scheme;
* Patients living more than 40 km from reference center;
* Patient depending on mechanical ventilation (more than 6 hours daily);
* Rapidly or reversible evolutive neuro-myopathy (Amyotrophic lateral sclerosis, Guillain Barré syndrome, myasthenia).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chronic respiratory failure due to neuromuscular diseases under non-invasive mechanical ventilation
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2024-03-08 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Gradation of quality of recorded signals at home | at day 1
  Expressed in number of readable signals for which the readability will be expressed in % of record time.

CONTACTS AND LOCATIONS:
Overall Officials: Frédéric Lofaso, MD, PhD, Principal Investigator — Department of physiology and functional explorations - Raymond Poincaré Hospital - APHP; Hélène Prigent, MD, PhD, Study Director — Department of physiology and functional explorations - Raymond Poincaré Hospital - APHP
Locations (1):
- Department of physiology and functional explorations - Raymond Poincaré Hospital - APHP, Garches, France

IPD SHARING:
Plan to Share IPD: No